CLINICAL TRIAL: NCT07071935
Title: A Pilot Randomized Clinical Trial of Early Ventilation in Amyotrophic Lateral Sclerosis (EVENT ALS)
Brief Title: A Clinical Trial of Early Ventilation in Amyotrophic Lateral Sclerosis (EVENT ALS)
Acronym: EVENT ALS
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, Jason Ackrivo, Assistant Professor of Medicine and Neurology, University of Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 858612; HT9425-25-1-0154 (Other Grant/Funding Number: Department of Defense)
Record Dates: First submitted 2025-07-08; First posted 2025-07-17 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Amyotrophic Lateral Sclerosis (ALS); Chronic Respiratory Failure; Neuromuscular Disease Patients; Neuromuscular Disease; Respiratory Insufficiency; Respiratory Insufficiency Requiring Mechanical Ventilation; Positive Pressure Ventilation; Non-invasive Ventilation; Non-invasive Ventilation Support; Non-invasive Ventilatory Support
Keywords: chronic respiratory failure; chronic neuromuscular respiratory failure; non-invasive ventilation; amyotrophic lateral sclerosis
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis; Neuromuscular Diseases; Respiratory Insufficiency | interventions — Noninvasive Ventilation; Continuous Positive Airway Pressure

STUDY DESIGN:
Intervention Model Description: Pilot randomized clinical trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Early Non-invasive Ventilation (Experimental): Participants randomized to this arm will be assigned to start therapy with non-invasive ventilation.
  Interventions: Device: Non-invasive ventilation
- Usual care (No Intervention): Participants randomized to this arm will receive usual care for amyotrophic lateral sclerosis.

INTERVENTIONS:
Device: Non-invasive ventilation — Non-invasive ventilation will be started earlier than usual respiratory care guidelines for ALS in the United States.
  Other Names: non-invasive positive pressure ventilation; bilevel positive airway pressure
  Arms: Early Non-invasive Ventilation

SUMMARY:
Amyotrophic lateral sclerosis (ALS) is a disease that causes weakness of the muscles of the body. The disease can eventually lead to severe breathing problems, which is the most common cause of death from ALS. The treatment for breathing is non-invasive ventilation (NIV). It is a machine that helps a person breathe by pushing air in and out of their lungs through a mask worn over the face. Research has shown that NIV can improve the quality of life and survival of someone with ALS. Unfortunately, NIV is not equally beneficial for everyone. The investigators do not yet know the best time or method for starting NIV in ALS. Europe and Canada allow starting NIV much earlier in ALS than the United States. Current recommendations for starting NIV are based on the opinion of experts rather than large research studies. Medical insurance companies will not cover NIV until significant breathing weakness occurs. After NIV is started, there is no evidence-based guidance on the best way to adjust NIV to benefit patients as much as possible. Some patients have difficulty tolerating NIV, but it is not clear how to identify these individuals ahead of time.

The investigators have created a new prediction tool that can identify patients at high risk of breathing problems within the next 6 months. This may help the study team identify who is more likely to benefit from starting NIV early. The investigators have published a paper that shows that NIV helps people with ALS live longer. This paper also showed that patients get more benefit with use NIV for at least 4 hours per day. The investigators published another paper that measured a gas called carbon dioxide (CO2), which goes high if someone's breathing is weakened. This paper showed that patients with ALS may live longer when CO2 levels are lowered using NIV. The investigators also have data suggesting that certain characteristics may predict who is less likely to use NIV at least 4 hours per day.

In this study, the investigators will collect pilot data on starting early NIV in individuals with ALS who do not yet meet insurance criteria for covering NIV. The research team will first use their previously published prediction tool to identify patient risk. Then, subjects would be randomized to start early NIV or to usual care. The usual care group would eventually start NIV as would occur if the participants were not in the study.

The purpose of this study is to collect data to help the investigators plan a larger randomized clinical trial. This study has 4 objectives. First, the project aims to identify individuals who would benefit from earlier NIV. The research team will use the original prediction tool to identify risk of severe breathing problems within the next 6 months. Second, the project aims to show that it is feasible to start NIV early. Third, the project aims to gather data on the effect of randomization on symptoms, CO2 levels, and outcomes. Fourth, the project aims to identify traits that may make someone less likely to use NIV.

DETAILED DESCRIPTION:
Background: Amyotrophic lateral sclerosis (ALS) is a progressive neurodegenerative disease with high morbidity and universal mortality predominantly due to respiratory failure. Non-invasive ventilation (NIV) improves quality of life (QoL) and extends survival in ALS beyond any medication.1-3 However, the best timing for NIV initiation is based only on expert opinion.4,5 For example, clinicians in the United States initiate NIV much later than European or Canadian guidelines,4,6,7 as payers do not cover NIV until significant respiratory impairment occurs. While potentially beneficial, early NIV initiation could increase burden for patients due to mask intolerance, claustrophobia, and disturbed sleep, possibly negating any clinical benefit. Similarly, there are no surrogate endpoints to guide NIV settings and mask selection. Thus, clinicians employ generic approaches despite significant disease heterogeneity. Given the variable onset and progression of ALS, strategies for anticipating respiratory risk and personalizing NIV management are critical to maximize NIV benefit while reducing its burden.

The investigators' ultimate goal is to conduct Phase III multicenter clinical trials which investigate early NIV strategies to improve quality of life and survival in individuals with ALS. Before embarking on a large RCT of early NIV in ALS, it is necessary to collect pilot data on feasibility, effect sizes, and personal factors associated with NIV usage. The study team's prior work has developed a novel clinical prediction tool which can stratify ALS patients at presentation into high versus low risk of respiratory insufficiency within 6 months, capable of identifying an enriched subgroup suitable for an interventional study. The investigators have performed semi-structured interviews which suggest that ALS patients value being proactive about their respiratory care. The investigators have shown that improving transcutaneous carbon dioxide (CO2) levels is associated with improved survival in ALS, suggesting that transcutaneous CO2 could be a surrogate endpoint for guiding NIV management. The investigators also have found that factors at time of NIV initiation, such as ALSFRS-R speech and dyspnea scores, are significantly associated with NIV adherence.

Clinical Intervention: In this RCT of patients who have yet to meet insurance criteria for NIV coverage, the research team will randomize individuals to early NIV versus usual care, stratified by 6-month risk of respiratory insufficiency as determined by the investigators' previously published novel clinical prediction tool.

Objective(s): The objectives in this pilot study are to collect: 1) feasibility data on randomization to early NIV; 2) estimates of effect sizes of early NIV versus usual care on endpoints such as QoL, transcutaneous CO2, symptoms, and survival; and 3) identify factors present at time of NIV initiation which predispose to low hourly usage of NIV. The research team will analyze results across randomization groups, as well as assess the interaction between randomization and predicted risk of respiratory insufficiency.

Study Design: This study will be a 3-center phase II pilot randomized clinical trial of incident ALS patients diagnosed in the last 6 months.

Clinical Impact: The proposed study will help the investigators understand the feasibility and safety of starting early NIV in ALS. The study team will assess effect sizes on clinical endpoints, which will be critical for planning a future large RCT. Lastly, the study team will learn about patient characteristics that may predispose to lower NIV adherence. The investigators will examine results across randomization and the interaction with predicted risk of respiratory insufficiency. Leveraging the clinical prediction tool may help identify an enriched patient population suitable for future interventional studies.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with ALS using the Gold Coast Criteria within the last 6 months
* Age ≥18 years
* Willingness and ability to participate in study procedures
* Provision of signed and dated informed consent form

Exclusion Criteria:

1. Current or prior or recommended/prescribed use of NIV including:

   i) bi-level positive pressure ventilation, such as a respiratory assist device or home ventilator ii) Current or prior use of continuous positive airway pressure, or "CPAP" therapy
2. Forced vital capacity <50% of predicted normal
3. Maximal inspiratory pressure > -60 cmH2O (eg, -50 or -40 cmH2O would be excluded)
4. Chronic use of supplemental oxygen at any part of the day
5. Enrollment in hospice
6. Current tracheostomy
7. Prior history of sleep apnea where non-invasive ventilation was used or recommended
8. Thoracic, abdominal, facial or ophthalmic surgery in the prior 6 weeks
9. Coughing up blood
10. Myocardial infarction in the previous 4 weeks
11. Absolute contraindication to NIV, which includes lethargy, obtundation, facial fractures, active pneumothorax, and airway obstruction (such as a tumor)
12. Presence of cognitive dysfunction that would impair ability to complete study procedures, as determined by neurology attending physician

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2029-05 (Estimated); Study Completion 2029-05 (Estimated)

PRIMARY OUTCOMES:
Time to first use of non-invasive ventilation | From enrollment to end of follow-up at approximately 1 year
  Number of days between randomization to first recorded overnight usage of non-invasive ventilation according to ventilation device data download.

SECONDARY OUTCOMES:
Quality of life questionnaire | From enrollment to completion of follow-up at approximately 1 year
  Quality of life will be measured by the ALS Specific Quality of Life questionnaire - short form (ALSSQOL-SF), a validated questionnaire to assess quality of life in terms applicable to a person with ALS. The questionnaire includes 20 questions scored on a scale of 0-10.
Transcutaneous carbon dioxide | From enrollment to end of follow-up at approximately 1 year
  Measured during the day in clinic using a transcutaneous carbon dioxide monitor. Units are in mmHg
Oxygen saturation using pulse oximetry | From enrollment to completion of follow-up at approximately 1 year
  Pulse oximeter used during the day during a clinic visit. Unites in % of saturated hemoglobin.
Epworth Sleepiness Scale - Alternative (ESS-ALT) questionnaire | From enrollment to completion of follow-up at approximately 1 year.
  The ESS-ALT includes 8 questions on likelihood of falling asleep during various activities and was designed for individuals with physical disabilities. Each question is rated on an ordinal integer scale of 0 (never) to 3 (high).
ALS Functional Rating Scale - Revised (ALSFRS-R) scores | From enrollment to completion of follow-up at approximately 1 year.
  The ALSFRS-R is a 12-item standardized questionnaire to assess the motor function status of an individual with ALS. Each of the 12 components of the questionnaire are scored on a scale of 0 to 4, with 4 being normal/no symptoms at all and 0 being severely symptomatic with little or no function.
Karolinska Sleepiness Scale (KSS) | From enrollment to completion of follow-up at approximately 1 year.
  The KSS questionnaire includes 1 question that is a 9-point ordinal integer scale asking the sleepiness level in the immediately preceding 10 minutes. The scale ranges from 1 (extremely alert) to 9 (very sleepy, great effort to keep awake, fighting sleep).
Global rate of change of breathing questionnaire | From enrollment to completion of follow-up at approximately 1 year.
  The global rate of change score for breathing will obtain a participant's subjective sense of their breathing status. The global rate of change score for the breathing will ask patients how their breathing is today by rating it on a Likert scale from -7 (extremely impaired) to +7 (extremely strong).
Global rate of change of sleep quality | From enrollment to completion of follow-up at approximately 1 year.
  The global rate of change score for sleep quality will obtain a participant's subjective sense of their sleep quality. The global rate of change score for the sleep quality will ask patients how their sleep quality is today by rating it on a Likert scale from -7 (extremely poor) to +7 (extremely good).
Tracheostomy-free survival time | Time in days between enrollment and either study withdrawal, death, placement of a tracheostomy, or completion of follow-up at approximately 1 year.
  Number of days between enrollment and the end of follow up, study withdrawal, or death without interval placement of a tracheostomy.
Hospitalizations | From enrollment to completion of follow-up at approximately 1 year.
  Number and time to hospitalizations during follow-up.
Average daily hourly usage of NIV | Between enrollment and completion of follow-up at approximately 1 year.
  This will be collected on subjects who are prescribed NIV within either study arm. Defined using telemonitoring portal data downloads (such as ResMed AirView for ResMed devices) which summarize average daily hourly usage over various specified time interval (e.g., the previous 30 days).
Vital capacity | From enrollment to completion of follow-up at approximately 1 year.
  Measured by performing a spirometry maneuver for vital capacity using a hand-held clinical-research grade spirometer in the sitting and upright position. Units are in liters.
Maximal inspiratory pressure | From enrollment to completion of follow-up at approximately 1 year.
  Measured using a hand-held digital manometer with the patient in the sitting and upright position.

CONTACTS AND LOCATIONS:
Overall Officials: Jason T Ackrivo, MD, MSCE, Principal Investigator — Perelman School of Medicine at the University of Pennsylvania
Locations (3):
- United States (3):
  - Penn State Hershey ALS Clinic, Hershey, Pennsylvania
  - Penn Comprehensive ALS Center at Pennsylvania Hospital, Philadelphia, Pennsylvania
  - Thomas Jefferson University Weinberg ALS Center, Philadelphi, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
Data dictionary and de-identified dataset
Supporting Information: Study Protocol, ICF, Analytic Code
Time Frame: Upon study completion and for up to 3 years after study end date.
Access Criteria: De-identified data available upon completion of a data sharing agreement

REFERENCES:
- [Background] Sarasate M, Gonzalez N, Cordoba-Izquierdo A, Prats E, Gonzalez-Moro JMR, Marti S, Lujan M, Calle M, Anton A, Povedano M, Farrero E. Impact of Early Non-Invasive Ventilation in Amyotrophic Lateral Sclerosis: A multicenter Randomized Controlled Trial. J Neuromuscul Dis. 2023;10(4):627-637. doi: 10.3233/JND-221658. PMID 37212068
- [Background] Gruis KL, Brown DL, Weatherwax KJ, Feldman EL, Chervin RD. Evaluation of sham non-invasive ventilation for randomized, controlled trials in ALS. Amyotroph Lateral Scler. 2006 Jun;7(2):96-9. doi: 10.1080/14660820600640604. PMID 16753973
- [Background] Ackrivo J, Hansen-Flaschen J, Wileyto EP, Schwab RJ, Elman L, Kawut SM. Development of a prognostic model of respiratory insufficiency or death in amyotrophic lateral sclerosis. Eur Respir J. 2019 Apr 18;53(4):1802237. doi: 10.1183/13993003.02237-2018. Print 2019 Apr. PMID 30728207
- [Background] Ackrivo J, Hsu JY, Hansen-Flaschen J, Elman L, Kawut SM. Noninvasive Ventilation Use Is Associated with Better Survival in Amyotrophic Lateral Sclerosis. Ann Am Thorac Soc. 2021 Mar;18(3):486-494. doi: 10.1513/AnnalsATS.202002-169OC. PMID 32946280